CLINICAL TRIAL: NCT00006092
Title: A Phase II Study of Arsenic Trioxide for Induction Therapy of Adult Patients With Relapsed or Refractory Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia and Previously Untreated Chronic Myeloid Leukemia With Blast Crisis
Brief Title: Arsenic Trioxide for Induction Therapy of Adult Patients With Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12395; NCI-1230 (Other: NCI)
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; lymphoid leukemia; myeloid and monocytic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphoid; Leukemia, Monocytic, Acute | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arsenic Trioxide Treatment (Experimental): Patients receive arsenic trioxide IV over 2-3 hours daily for 28 days. Patients who respond may receive a second course of therapy beginning 28 days from the last dose of the first course.
  Interventions: Drug: Arsenic Trioxide

INTERVENTIONS:
Drug: Arsenic Trioxide
  Other Names: Trisenox

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have recurrent or refractory acute lymphoblastic leukemia or chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the rate of clinical and hematologic response in patients with Philadelphia chromosome-positive recurrent or refractory acute lymphoblastic leukemia or previously untreated or recurrent or refractory blastic phase chronic myelogenous leukemia when treated with arsenic trioxide.
* Determine the duration of hematologic response and overall survival of these patients when treated with this regimen.
* Determine the pattern of clinical adverse experience in these patients when treated with this regimen.
* Determine the pharmacokinetic profile of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive arsenic trioxide IV over 2-3 hours daily for 28 days. Patients who respond may receive a second course of therapy beginning 28 days from the last dose of the first course.

Patients are followed monthly for 3 months, every 2 months for 6 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 24-49 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Acute lymphoblastic leukemia

    * Philadelphia chromosome (Bcr-abl) positive
    * Refractory to initial therapy OR recurrent following 1 induction therapy regimen with or without consolidation therapy and/or bone marrow transplantation
  * Blastic phase chronic myelogenous leukemia

    * Philadelphia chromosome (Bcr-abl) positive
    * Previously untreated OR recurrent or refractory following 1 induction therapy regimen with or without consolidation therapy including imatinib mesylate
* Must not be eligible for bone marrow transplant

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 times upper limit of normal (ULN)
* AST/ALT no greater than 2 times ULN

Renal:

* Creatinine no greater than 2.0 times ULN
* Creatinine clearance greater than 70 mL/min

Cardiovascular:

* No uncontrolled angina
* No New York Heart Association class III or IV heart disease
* No second degree heart block without pacemaker

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* HIV negative
* No uncontrolled infection or other serious concurrent illness
* No peripheral neuropathy
* No potassium less than 3.0 or greater than 5.5 mEq/L that can not be corrected OR
* No magnesium less than 1.2 or greater than 2.5 mEq/L that can not be corrected
* Electrolyte imbalances must be corrected prior to study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* At least 28 days since prior chemotherapy
* At least 24 hours since prior hydroxyurea
* No prior arsenic trioxide
* No other concurrent cytotoxic chemotherapy except intrathecal chemotherapy for CNS leukemia

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 28 days since prior radiotherapy
* No concurrent radiotherapy including for palliation

Surgery:

* Not specified

Other:

* At least 14 days since prior imatinib mesylate
* No other concurrent investigational agents
* No concurrent amphotericin B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2000-08; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Objective Rate of Response (ORR) | 2.5 years
  Determine the rate of clinical and hematologic response in patients with Philadelphia chromosome-positive recurrent or refractory acute lymphoblastic leukemia or previously untreated or recurrent or refractory blastic phase chronic myelogenous leukemia when treated with arsenic trioxide.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P. Loughran, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States